CLINICAL TRIAL: NCT07158827
Title: Expanded Access to Tavapadon
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C25-978
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme; Parkinson Disease; Tavapadon; ABBV-1751; C25-978
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tavapadon — Oral: Tablet

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to tavapadon prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=C25-978